CLINICAL TRIAL: NCT03008473
Title: Placement of the Uniblocker Under the Guidence of Chest Computerized Tomography
Brief Title: Chest CT for the Placement of the Uniblocker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 20161229
Record Dates: First submitted 2016-12-29; First posted 2017-01-02 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2016-12

CONDITIONS: Therapeutic Procedural Complication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- video laryngoscope and chest CT iminge (Experimental): First,the operator calculate the distance between the carina and the glottis by CT image and make a marker on the Uniblocker. Then the operator inserted the Uniblocker into the trachea and advanced toward the left main-stem bronchus via the video laryngoscope untill see marker just at the glottis then stopped the insertion .Second, a single lumen tube with appropriate size was intubated via video laryngoscope into the appropriate depth.Third,the Fiberoptic bronchoscopy(FOB) was inserted into single lumen tube to assess the position of the Uniblocker and the injuries of bronchi and carina
  Interventions: Device: video laryngoscope and chest CT iminge
- Conventional intubation of Uniblocker (Experimental): First, a conventional single lumen tube (SLT) was inserted into trachea at optimal depth via video laryngoscope. Second, a Uniblocker was inserted through SLT and directed to the left main-stem bronchus. Third, an FOB was inserted into the SLT to adjust the Uniblocker to optimal position and assessed the injuries of bronchi and carina.
  Interventions: Device: Conventional intubation of uniblocker

INTERVENTIONS:
Device: video laryngoscope and chest CT iminge
  Arms: video laryngoscope and chest CT iminge
Device: Conventional intubation of uniblocker
  Arms: Conventional intubation of Uniblocker

SUMMARY:
Video laryngoscope and chest CT iminge for the placement of the Uniblocker

DETAILED DESCRIPTION:
Comparing the traditional method of Uniblocker intubation and video laryngoscope combined with chest CT iminge guide the precise localization of Uniblocker

ELIGIBILITY:
Inclusion Criteria:

BMI less than 35 kg/m2 ASA classifications of I-III, Modified Mallampati classification 1 or 2 Under general anesthesia

Exclusion Criteria:

* Age younger than 18 yr or older than 65 yr
* ASA class IV or V
* Abnormalities of the heart, brain, liver, lung, kidney and coagulation functions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-09-24 (Actual); Study Completion 2017-09-24 (Actual)

PRIMARY OUTCOMES:
Intubation Time | 5min

CONTACTS AND LOCATIONS:
Overall Officials: Ximing Qi, PHD, Study Director — The First Hospital of Qinhuangdao
Locations (1):
- The first hospital of Qinhuangdao, Qinhuangdao, Hebei, China

IPD SHARING:
Plan to Share IPD: Yes